CLINICAL TRIAL: NCT06548308
Title: Comparison of Corneal Incision Versus Toric Intraocular Lens Techniques Used in Cataract Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/734
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Cataract Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corneal Incision (Experimental)
  Interventions: Diagnostic Test: Corneal Incision
- Toric Intraocular (Active Comparator)
  Interventions: Other: Toric Intraocular

INTERVENTIONS:
Diagnostic Test: Corneal Incision — Astigmatism will be assessed by objective and subjective refraction by using the Autorefrectometer and retinoscop.Autorefrectometer uses to acsess the refracive state of eye by which we measure the astigmatim in patients eyes .Then after ctaract surgry in the next followup we will again use autorefrectometer to take readings and these both will be compared on visits among patients undergoing two procedures.
  Arms: Corneal Incision
Other: Toric Intraocular — Two cataract surgery techniques will be used .1 : Toric IOL lenses designed with a unique shape to help provide clear vision at all distances for individuals with astigmatism compared to give better results specially in astigmatic patients.2: Corneal Inscion is which eye surgeon makes a very small opening on the eye, next to the outer corner. to remove the catract during surgry .
  Arms: Toric Intraocular

SUMMARY:
Eyesight and quality of life improves in patients after refractive cataract surgery because this surgery treats myopia, hyperopia and presbyopia except astigmatism. In order to make a patient spectacle free Ophthalmologists use different methods during cataract surgery to minimize astigmatism.

DETAILED DESCRIPTION:
These methods includes limbal relaxing incisions (LRIs) or the insertion of toric IOLs, which are specifically intended to cancel out pre-existing astigmatism and astigmatic keratometry. This research will be conducted to see which method benefits more for treating preoperative astigmatism in eye.

ELIGIBILITY:
Inclusion Criteria:

* Both genders were included.
* Patients having astigmatism was included. Patients having cataract was included.
* Eyes having no other ocular pathology was included.
* Patients having no history of corneal scar was included

Exclusion Criteria:

* Eyes having any ocular pathology will be excluded.
* Patients with corneal suture will be excluded.
* Those using contact lenses instead of spectacles for vision correction will be excluded.
* Participants with a history of eye surgery within the past year will be excluded.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
postoperative visual acuity | 12 Months
  The postoperative visual acuity and refractive outcomes between patients undergoing cataract surgery with corneal incision and those with toric IOL implantation.
effectiveness of astigmatism correction | 12 months
  Investigate the effectiveness of astigmatism correction achieved by both toric iol and corneal inscion technique and determine the degree of residual astigmatism in both groups after followups .

CONTACTS AND LOCATIONS:
Locations (1):
- Zubaida eyecare center sabzazar, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No